CLINICAL TRIAL: NCT04267224
Title: Efficacy and Safety of Early Versus Late Loading Dose of Ticagrelol in Patients With ST Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Early Versus Late Loading of Ticagrelol in Patients With STEMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hany Rayek Maher, Resident doctor, Assiut University
Other Study IDs: Ticagrelor in STEMI patients
Record Dates: First submitted 2019-09-25; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early group: Patients receiving the loading dose of Ticagrelol 90 mg more than 60 minutes before PCI.
  Interventions: Drug: Ticagrelor 90mg
- Late group: Patients receiving the loading dose of Ticagrelol 90 mg less than 60 minutes before PCI.
  Interventions: Drug: Ticagrelor 90mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — Ticagrelor is a direct-acting inhibitor of the platelet P2Y12 receptor with a rapid antiplatelet effect. It has been shown to reduce the rate of major cardiovascular events among patients with acute coronary syndromes, as compared with Clopidogrel, and has the potential to improve coronary reperfusion and the prognosis for patients with STEMI treated with primary PCI.
  Other Names: Early versus late loading with Ticagrelol

SUMMARY:
Current guidelines recommend percutaneous coronary intervention (PCI) for most patients with ST segment elevation acute myocardial infarction (STEMI) or with non ST segment elevation acute coronary syndrome (NSTEACS) . In STEMI patients, PCI is advised in all patients in the first 12 hours after onset of symptoms, the earlier the better.

This condition is referred to as "no-reflow phenomenon." , no-reflow is defined as suboptimal myocardial reperfusion through a part of coronary circulation without angiographic evidence of mechanical vessel obstruction.

Effective antiplatelet therapy combining the inhibition of both thromboxane A2-dependent platelet aggregation and P2Y12 receptors is necessary in patients undergoing percutaneous coronary intervention (PCI), particularly those with ST-segment elevation myocardial infarction (STEMI).

The goal of DAPT (Aspirin and P2Y12 receptor inhibitors) is to reduce the risk of ischemic events such as (re)-infarction and the risk of stent thrombosis after PCI. It is logical to assume that early administration of a P2Y12 inhibitor prior to PCI (referred to as pre-treatment) should provide greater benefit given the fact that even the fastest acting oral P2Y12 inhibitors take at least 30-60 min.

Various studies and meta-analyses suggested that pretreatment with Clopidogrel in patients with STEMI could reduce the rate of ischemic events without excess bleeding, but its effectiveness may be limited by its slow onset of action and the variable response. In contrast, the new oral P2Y12-receptor antagonists (Prasugrel or Ticagrelol) inhibit platelet function in less than 1 hour, which is compatible with transfer times for primary PCI.

Ticagrelor is a direct-acting inhibitor of the platelet P2Y12 receptor with a rapid antiplatelet effect. It has been shown to reduce the rate of major cardiovascular events among patients with acute coronary syndromes, as compared with Clopidogrel, and has the potential to improve coronary reperfusion and the prognosis for patients with STEMI treated with primary PCI. but The issue of pre-treatment with ticagrelor for patients with STEMI remains an area of ongoing debate; whether they are initiated in the pre-hospital setting, emergency department, or anywhere .

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed as STEMI according to criteria developed by the European Society of Cardiology.
2. Onset of maximal intensity of chest pain within 12 hours before procedure.

Exclusion Criteria:

1. Contraindication to Ticagrelor (e.g., hypersensitivity, active bleeding, history of previous intracranial hemorrage, moderate to severe hepatic impairment, GI bleeding within the past 6 months, major surgery within past 4 weeks)
2. Patient who has recently received loading dose of Clopidogrel or are on chronic treatment of Clopidogrel.
3. Patients who are on oral anticoagulation therapy that cannot be stopped (i.e., patient with prosthetic valves, chronic AF…etc)
4. Patients with clinically significant thrombocytopenia.
5. Previous enrolment in the present study (Upstream use of GPIIb/IIIa is not recommended as a concomitant treatment)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include 800 patients (divided in 2 groups), 400 patients receiving the loading dose early more than 60 minutes before the procedure and 400 patients receiving the loading dose in late less than 60 minutes before the procedure.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of Major adverse cardiovascular events (MACE) | 6 weeks
  Efficacy end point
The occurrence of major or minor bleeding | 6 weeks
  safety endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Hany R. Maher, Principal Investigator — Assiut University